CLINICAL TRIAL: NCT04553757
Title: Seizure Control as a New Metric in Assessing Efficacy of Tumor Treatment in Patients With Low Grade Glioma
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-0124; NCI-2020-06510 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0124 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Brain Neoplasm; Low Grade Glioma; Seizure Disorder
MeSH Terms: conditions — Brain Neoplasms; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (survey): Patients complete a seizure assessment survey over 5 minutes at each clinic visit.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Complete survey

SUMMARY:
This study investigates how seizures can vary over time with changes in low grade gliomas and its treatments. This study may help doctors find symptoms or triggers of seizures earlier than normal, and ultimately earlier care or treatment for seizures.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the rate of change of seizure frequency and the status of the tumor at each data collection point.

SECONDARY OBJECTIVES:

I. To obtain sufficient number of patients' data in order to power the analysis to determine whether a change in seizure frequency correlates with tumor control.

II. Evaluate progression free survival and overall survival when compared with seizure control.

OUTLINE:

Patients complete a seizure assessment survey over 5 minutes at each clinic visit.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Primary brain tumors (separated by World Health Organization [WHO] grade I-IV)
* History of seizures secondary to brain tumor
* On tumor directed treatment
* Magnetic resonance imaging (MRI) within 2 weeks of clinic visit where seizure assessment takes place

Exclusion Criteria:

* Patients without seizures
* Patients with intracranial lesions other than primary brain tumor
* Patients not undergoing tumor directed treatment
* Absence of recent (within 2 weeks) MRI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with primary brain tumors with a history of seizures secondary to brain tumor.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of change of seizure frequency | Baseline to 2 years
  Both average composite scores as well as individual question scores from the seizure survey will be evaluated. Will perform descriptive statistics to characterize the demographic and disease-related features of this population. Will perform regression analyses to the relationship of survey results to clinical and radiographic features. Cox regression analyses for other relevant post-hoc analyses may be performed.
Status of tumor | Up to 2 years
  Radiographic information will be derived from brain MRIs performed on each patient at time of diagnosis, and subsequently at times of survey administration. Will perform descriptive statistics to characterize the demographic and disease-related features of this population. Will perform regression analyses to the relationship of survey results to clinical and radiographic features. Cox regression analyses for other relevant post-hoc analyses may be performed.

SECONDARY OUTCOMES:
Patient data collection | Up to 2 years
  Will obtain sufficient number of patients' data in order to power the analysis to determine whether a change in seizure frequency correlates with tumor control. Clinical information to be extracted from the medical record includes but not limited to; date of birth, gender, date of diagnosis, clinical symptoms referable to the brain tumor, functional status and age at diagnosis, treatments applied, dates of progression, and date of death. Radiographic information will be derived from brain MRIs performed on each patient at time of diagnosis, and subsequently at times of survey administration. Will perform descriptive statistics to characterize the demographic and disease-related features of this population.
Progression-free survival (PFS) | Up to 2 years
  Will evaluate PFS when compared with seizure control.
Overall survival (OS) | Up to 2 years
  Will evaluate OS when compared with seizure control.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Aaroe, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org